CLINICAL TRIAL: NCT04114552
Title: Follow up of Patients After a Visit to Tourcoing Emergency Department for an Ankle Sprain
Acronym: CHEVILLE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RNI_2019_23; 2019-A01824-53 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Ankle Sprains
Keywords: inversion trauma; Ankle sprain; physical examination; therapy; recurrence
MeSH Terms: conditions — Ankle Injuries; Recurrence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires — 6 weeks after the trauma,during the call, an oral questionnaire will be proposed to collect data on patients' management since they have left the emergency department.
  After the call, socio-demographic characteristics, trauma mechanism, medics management will be extracted from the patient's medical records

SUMMARY:
Ankle sprain is very common. In France, its daily incidence is estimated at 6000. It often causes pain, a temporary period of disability and can results in recurrence and chronic ankle instability. Therefore, an early management and follow up treatment is necessary. Now, functional treatment is clinically the treatment strategy of choice for ankle sprain. It is based on rest, ice, compression, elevation and can use a functional support (like an ankle brace). To evaluate gravity and improve management, a clinical assessment delayed between 4 and 5 days post injury is necessary.

ELIGIBILITY:
Inclusion Criteria:

Consulted for ankle trauma as primary reason Agreeing to participate in the telephone survey 6 weeks after trauma Affiliation in a social security scheme

Exclusion Criteria:

Patients deprived of liberty Patients with an unbalanced psychiatric disease If consultation delayed 48 hours due to trauma Patients with fracture Patients with Chopart or Lisfranc injury Pregnant women People who do not speak French

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who consulted at Tourcoing emergency department for an ankle sprain
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Rate of patients who received a five days post injury new clinical assessment | at 6 weeks

SECONDARY OUTCOMES:
Oral questionnaires | At 6 weeks
  The questionnaire will ask questions around their socio-demographic characteristics, trauma mechanism, medics management since they have left the emergency department.
Rate of patients receiving physiotherapy | At 6 weeks
Rate of patients with recurrence | At 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hacène MOUSSOUNI, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Ch Tourcoing, Tourcoing, France